CLINICAL TRIAL: NCT05100771
Title: Volumétrie Optimisée en Radiologie : intérêt en IRM Cérébrale pédiatrique Dans l'Exploration de l'épilepsie Focale
Brief Title: Optimized Volumetry in Radiology: Interest in Pediatric Brain MRI in the Exploration of Focal Epilepsy
Acronym: ORACLE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR210107
Record Dates: First submitted 2021-09-28; First posted 2021-10-29 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Focal Epilepsy
Keywords: Brain MRI; Radiology; Pediatry
MeSH Terms: conditions — Epilepsies, Partial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental group: The experimental group will be made up of patients with focal epilepsy
  Interventions: Other: Pediatric brain MRI

INTERVENTIONS:
Other: Pediatric brain MRI — Routine brain MRI with automated quantitative information (brain volumetry and T1 relaxometry)

SUMMARY:
Multicentre cross-sectional study with prospective recruitment comparing the detection rate of lesions on brain MRI without and with quantitative volumetry and T1 relaxometry information during the management of children with suspected focal epilepsy.

DETAILED DESCRIPTION:
Focal epilepsies are a very heterogeneous group comprising epilepsies of structural, genetic, metabolic, immune and infectious etiologies. In daily practice, epilepsy is considered as structural if lesions are visible on brain MRI in a location consistent with electro-clinical data. In the absence of visible lesion and clinico-biological arguments for a genetic, metabolic, immune or infectious cause, these epilepsies can be divided into two groups: self-limited focal epilepsies (formerly called idiopathic or functional), such as benign epilepsy with centrotemporal spikes (SLECTS) and secondly epilepsies of unknown causes. This classification underlines the idea that a lesion might be responsible for the epileptic disease but could be invisible due to the lack of sensitivity of our current diagnostic methods, especially in imaging.

The prevalence of patients with non lesional epilepsy defined by MRI is significantly higher in children (31%) than in adults (21%). Epileptic patients with normal conventional MRI have a lower chance of having surgery than those with lesions demonstrated by presurgical MRI and, if so, less chance of becoming seizure-free. It can be challenging to depict brain volume abnormalities in the pediatric population on MRI. The major challenge is therefore to raise sensitivity of brain imaging analysis. Voxel-based morphometric MRI post-processing in MRI-negative epilepsies can be a practical and valuable tool to aid subtle MRI abnormalities detection and confirm visually identified questionable abnormalities in patients with focal epilepsy.

In this study, we prospectively included children with suspected focal epilepsy having a brain MRI using a MP2RAGE sequence and a post-processing morphometric analysis program (MAP) allowing us to obtain automatically both brain volumetry and T1 relaxometry. The MAP has been validated with reference ranges in healthy children. Our hypothesis was that the quantitative information will improve the sensitivity of brain MRI in children with suspected focal epilepsy. The objectives were to compare the rate of detection of a focal cerebral lesion on the brain MRI carried out during the exploration of suspected focal epilepsy without then with the quantitative volumetry and T1 relaxometry obtained in the inclusion center and then by double anonymized review.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 1-18 years
* Referred or followed by a pediatrician for epilepsy with focal onset
* Requiring brain MRI as part of the work-up

Exclusion Criteria:

* Opposition of the child and/or parent to data processing
* MRI not interpretable
* Clinical and epileptic data not available or not specifying focus

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All participants will be included in a visit as part of their routine follow-up with a pediatric epilepsy specialist for a work-up including clinical examination, EEG examination and assessment of symptomatology between clinical, EEG and MRI.
  All visits and examinations are part of routine care. Additional quantitative data from the MRI will not influence medical management in any way.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
rate of detection of a focal cerebral lesion on the brain MRI | Inclusion visit
  carried out during the exploration of suspected focal epilepsy without then with the quantitative volumetry and T1 relaxometry obtained in the inclusion center and then by double anonymized review

SECONDARY OUTCOMES:
Radiologist's confidence level in detecting lesions seen on MRI without the automated quantitative data | Inclusion visit
  Measured by a semi-quantitative visual analogue scale in the detection of brain lesions observed on MRI
Radiologist's confidence level in detecting lesions seen on MRI with the automated quantitative data | Inclusion visit
  Measured by a semi-quantitative visual analogue scale in the detection of brain lesions observed on MRI
pediatric brain MRIs interpretation without the additional quantitative brain information | Inclusion visit
  Inter-observer agreement in terms of normal or not normal MRI and in case of abnormality, the type of abnormality
pediatric brain MRIs interpretation with the additional quantitative brain information | Inclusion visit
  Inter-observer agreement in terms of normal or not normal MRI and in case of abnormality, the type of abnormality
Clinical examination | Inclusion visit
  Assessed by weight in kgs and height in cm, International League against epilepsy ( ILAE) classification
electroencephalography | Inclusion visit
  Assessed by focal abnormalities and area
Presentation of brain volumetry and T1 relaxometry in table form and map form | Inclusion visit
  pourcentage of choice between the table form and the map form depending on the radiologists

CONTACTS AND LOCATIONS:
Overall Officials: Baptiste Morel, Principal Investigator — CHU Tours
Locations (5):
- France (5):
  - CHU Angers, Angers
  - CHU Grenoble, Grenoble
  - CHU Montpellier, Montpellier
  - CHU Rennes, Rennes
  - Hôpital Clocheville, Tours

IPD SHARING:
Plan to Share IPD: Undecided